CLINICAL TRIAL: NCT00562978
Title: A Phase I/II Trial of Escalating Dose of Yttrium-90-labeled Anti-CD20 Monoclonal Antibody in Combination With High-Dose Etoposide and Cyclophosphamide Followed by AHSCT for Patients With Relapsed B-Cell Non-Hodgkin's Lymphoma
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan, Etoposide, Cyclophosphamide, and an AHSCT in Non-Hodgkin's Lymphoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 98153; P30CA033572 (NIH); P01CA030206 (NIH); CHNMC-98153; CDR0000574716 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent mantle cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell | interventions — Filgrastim; Cyclophosphamide; Etoposide; ibritumomab tiuxetan

ARMS (2):
- Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg (Experimental): * Preparation for AHSCT: Peripheral blood stem cells (PBSCs) are collected via leukapheresis. Samples are analyzed by cytogenetic studies, immunophenotyping, and gene rearrangement. Patients with an adequate number of collected CD34-positive cells (≥ 3 times 10^6 /kg) proceed to radioimmunotherapy.
  * Radioimmunotherapy: Patients receive yttrium Y 90 ibritumomab tiuxetan and undergo bone marrow biopsy and dose estimation.
  * Chemotherapy: Patients receive etoposide IV and cyclophosphamide IV
  * AHSCT: Patients undergo reinfusion of PBSCs.
  * Growth factor therapy: Patients receive filgrastim (G-CSF) IV. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: etoposide; Procedure: AHSCT; Radiation: yttrium Y 90 ibritumomab tiuxetan
- Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg (Experimental): * Preparation for AHSCT: Peripheral blood stem cells (PBSCs) are collected via leukapheresis. Samples are analyzed by cytogenetic studies, immunophenotyping, and gene rearrangement. Patients with an adequate number of collected CD34-positive cells (≥ 3 times 10^6 /kg) proceed to radioimmunotherapy.
  * Radioimmunotherapy: Patients receive yttrium Y 90 ibritumomab tiuxetan and undergo bone marrow biopsy and dose estimation.
  * Chemotherapy: Patients receive etoposide IV and cyclophosphamide IV
  * AHSCT: Patients undergo reinfusion of PBSCs.
  * Growth factor therapy: Patients receive filgrastim (G-CSF) IV. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: etoposide; Procedure: AHSCT; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
  Other Names: Cytoxan
Drug: etoposide
  Other Names: VP-16
Procedure: AHSCT
  Other Names: autologous hematopoietic stem cell transplantation
Radiation: yttrium Y 90 ibritumomab tiuxetan
  Other Names: Zevalin

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as etoposide and cyclophosphamide, work in different ways to kill cancer cells or stop them from growing. Giving radiolabeled monoclonal antibodies together with etoposide and cyclophosphamide before a peripheral blood stem cell transplant may be an effective treatment for non-Hodgkin lymphoma.

PURPOSE: This phase I/II trial is studying the side effects and best dose of yttrium Y 90 ibritumomab tiuxetan when given together with etoposide and cyclophosphamide followed by an autologous stem cell transplant and to see how well it works in treating patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the safety and efficacy of a new preparative regimen of yttrium Y 90 ibritumomab tiuxetan in combination with high-dose etoposide and cyclophosphamide followed by autologous stem cell transplantation (ASCT) for treatment of patients with poor-risk, relapsed, or refractory non-Hodgkin lymphoma (NHL).
* To determine the maximum tolerated dose of yttrium Y 90 ibritumomab tiuxetan which can be given with high-dose etoposide and high-dose cyclophosphamide followed by ASCT in patients with NHL.
* To perform dosimetry study to estimate the radiation dose delivered to the tumor and normal organs.
* To evaluate the short-term and long-term complications of this new preparative regimen.

OUTLINE: This is a phase I does-escalation study of yttrium Y 90 ibritumomab tiuxetan followed by an open-label phase II study.

* Preparation for transplantation: Peripheral blood stem cells (PBSCs) are collected via leukapheresis. Samples are analyzed by cytogenetic studies, immunophenotyping, and gene rearrangement. Patients with an adequate number of collected CD34-positive cells (≥ 3 times 10^6 /kg) proceed to radioimmunotherapy.
* Radioimmunotherapy: Patients receive yttrium Y 90 ibritumomab tiuxetan IV on days -21 and -14. Patients undergo bone marrow biopsy and dose estimation on day -7.
* Chemotherapy: Patients receive etoposide IV on day -4 and cyclophosphamide IV over 2 hours on day -2.
* Transplantation: Patients undergo reinfusion of PBSCs on day 1.
* Growth factor therapy: Patients receive filgrastim (G-CSF) IV beginning on day 1 and continuing until blood counts recover.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven diagnosis of low- or intermediate-grade* non-Hodgkin lymphoma (NHL) including any of the following:

  * Follicular small cleaved
  * Follicular mixed
  * Follicular large cell
  * Diffuse small cleaved
  * Diffuse mixed
  * Diffuse large cell
  * Immunoblastic (working formulation B, C, D, E, F, G and H) NOTE: *A new classification scheme for adult non-Hodgkin lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low-", "intermediate-", or "high-" grade lymphoma. However, this protocol uses the former terminology.
* Mantle cell and transformed low-grade lymphomas allowed
* Demonstrated monoclonal CD20-positive B-cell population in lymph nodes and/or bone marrow
* Favorable biodistribution on imaging dose
* Patient either relapsed after achieving a complete (CR) or partial response (PR) to prior therapy, never responded to prior therapy, or has poor-risk disease

  * Sensitivity of disease based on 1 of the following:

    * Induction failure: patients who did not achieve a CR or PR from induction chemotherapy
    * Resistant relapse: patients who did not achieve a CR or PR from the most recent standard salvage chemotherapy
    * Sensitive relapse: patients who did achieve a CR or PR from the most recent standard salvage chemotherapy
  * Poor-risk disease defined as any of the following:

    * Age-adjusted International Prognostic Index (IPI) High- (3 risk factors) or High-Intermediate (2 risk factors) based on the following risk factors:

      * Stage III-IV disease
      * Elevated serum lactate dehydrogenase level
      * ECOG performance status 2-4
    * Patients with aggressive NHL including mantle cell lymphoma and who required 2 different induction chemotherapy regimens to achieve a CR/PR
    * Patients with B-cell NHL and who failed to achieve a CR after adequate induction chemotherapy regimen(s)
* Patients must have bone marrow aspiration and biopsy within 42 days before salvage chemotherapy or stem cell collection which show ≤ 10% lymphomatous involvement of total cellularity
* Normal cytogenetic study on bone marrow (prior to salvage chemotherapy or stem cell collection)

  * Cytogenetic study on peripheral blood is acceptable if bone marrow biopsy has already been done and shows no sign of myelodysplastic syndrome (MDS) or lymphoma and a repeat bone marrow is deemed unnecessary by attending physician
* No active or prior history of CNS diseases
* No human anti-mouse antibody (HAMA) or human anti-chimeric antibody

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 or Karnofsky PS 80-100%
* Platelet count normal
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min
* FEV_1 > 65% of predicted or DLCO ≥ 50% of predicted
* LVEF > 50% by ECHO or MUGA scan
* Bilirubin ≤ 1.5 times normal
* SGOT or SGPT ≤ 2 times normal
* HIV antibody-negative
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinoma, or other cancer from which the patient has been disease-free for at least five years
* No active evidence of hepatitis B or C infection
* No hepatitis B surface antigen positivity
* No history of alcohol abuse
* Body weight ≤ 250 pounds

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients who have received involved field external beam therapy to area excluding lung, heart, liver and kidney are allowed, but will be evaluated on a case-by-case basis
* Patients must have recovered from last therapy and should be at least four weeks from prior radiation or chemotherapy
* No prior radioimmunotherapy
* No prior bone marrow transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2000-05-16 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Auayporn P. Nademanee, MD, Study Chair — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg; Zevalin 1000 cGy + VP-16 60 mg/kg +: * Preparation for AHSCT: Peripheral blood stem cells (PBSCs) are collected via leukapheresis. Samples are analyzed by cytogenetic studies, immunophenotyping, and gene rearrangement. Patients with an adequate number of collected CD34-positive cells (≥ 3 times 10^6 /kg) proceed to radioimmunotherapy.
  * Radioimmunotherapy: Patients receive yttrium Y 90 ibritumomab tiuxetan and undergo bone marrow biopsy and dose estimation.
  * Chemotherapy: Patients receive etoposide IV and cyclophosphamide IV
  * AHSCT: Patients undergo reinfusion of PBSCs.
  * Growth factor therapy: Patients receive filgrastim (G-CSF) IV. Treatment continues in the absence of disease progression or unacceptable toxicity.
  filgrastim
  cyclophosphamide
  etoposide
  AHSCT
  yttrium Y 90 ibritumomab tiuxetan
Period: Overall Study
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg +
Started | 6 | 48
Completed | 5 | 37
Not Completed | 1 | 11
Not completed — Patient had imaging dose only | 1 | 11

BASELINE CHARACTERISTICS:
Groups:
- Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg: * Preparation for AHSCT: Peripheral blood stem cells (PBSCs) are collected via leukapheresis. Samples are analyzed by cytogenetic studies, immunophenotyping, and gene rearrangement. Patients with an adequate number of collected CD34-positive cells (≥ 3 times 10^6 /kg) proceed to radioimmunotherapy.
  * Radioimmunotherapy: Patients receive yttrium Y 90 ibritumomab tiuxetan and undergo bone marrow biopsy and dose estimation.
  * Chemotherapy: Patients receive etoposide IV and cyclophosphamide IV
  * AHSCT: Patients undergo reinfusion of PBSCs.
  * Growth factor therapy: Patients receive filgrastim (G-CSF) IV. Treatment continues in the absence of disease progression or unacceptable toxicity.
  filgrastim
  cyclophosphamide
  etoposide
  AHSCT
  yttrium Y 90 ibritumomab tiuxetan
- Total: Total of all reporting groups
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg | Total
Number analyzed (Participants) | 6 | 48 | 54
Age, Continuous [Median (Full Range); unit: Years] | 54 [39 to 59] | 50 [23 to 59] | 50 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 20 | 21
  Male | 5 | 28 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 43 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 48 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete Response (CR)
Description: Complete response is defined as complete disappearance of all measureable evidence of non-evaluable disease. No new lesions. No disease related symptoms. No evidence of non-evaluable disease, including normalization of markers and other abnormal lab values. All measureable, evaluable and non-evaluable lesions and sites must be assessed using the same techniques as baseline.
Time Frame: Assessed up to 5 years post-ASCT
Population: Patients had favorable bio-distribution on imaging dose and received the study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg: Zevalin to deliver 1000 cGy highest normal organ excluding spleen and bone marrow with VP-16 40 mg/kg and Cytoxan 100 mg/kg. Patients underwent therapy on day -14 with VP-16 given on day -4, Cytoxan given on day -2 and PBSC infused on day +1.
- Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg: Zevalin to deliver 1000 cGy highest normal organ excluding spleen and bone marrow with VP-16 60 mg/kg and Cytoxan 100 mg/kg. Patients underwent therapy on day -14 with VP-16 given on day -4, Cytoxan given on day -2 and PBSC infused on day +1.
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg
Number analyzed (Participants) | 5 | 37
Participants | 4 | 32

2. Primary Outcome: Number of Patients With Grade 3 or Greater Toxicity
Description: The NCI Common Toxicity Criteria (CTC Version 2.0) are used. The patients, whose toxicities are grade 3 or greater and at possibly related to the study treatment, are reported.
Time Frame: From initial of study treatment to Day 100 post-ASCT
Population: Patients had favorable bio-distribution on imaging dose and received the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg
Number analyzed (Participants) | 5 | 37
Participants | 5 | 37

3. Primary Outcome: 5-Year Overall Survival (Phase II)
Description: Overall survival (OS) was measured from peripheral stem cell infusion to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula. [Breslow NE, Day NE. Statistical methods in cancer research: volume II, the design and analysis of cohort studies. IARC Sci Publ 1987;82:1-406.]
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to death due to any cause, assessed up to 5 years
Population: Patients had favorable bio-distribution on imaging dose and received the study treatment
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg
Number analyzed (Participants) | 5 | 37
percentage of probability | 60 [13 to 88] | 86 [71 to 94]

4. Primary Outcome: 5-Year Disease-free Survival (Phase II)
Description: Disease-free survival (DFS) was defined as time from peripheral stem cell infusion to relapse or death. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works. Disease-free survival was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula [Breslow NE, Day NE. Statistical methods in cancer research: volume II, the design and analysis of cohort studies. IARC Sci Publ 1987;82:1-406.]
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to first observation of relapse or death due to any cause, whichever comes first, assessed up to 5 years
Population: Patients had favorable bio-distribution on imaging dose and received the study treatment
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg
Number analyzed (Participants) | 5 | 37
percentage of probability | 60 [13 to 88] | 62 [45 to 76]

ADVERSE EVENTS:
Time Frame: Adverse Event and Vital Status data both were captured from the initial treatment to the off protocol, up to 5 years.
Description: Among the 54 enrolled patients, 12 patients had unfavorable bio-distribution on imaging dose. Those 12 patients didn't receive any study drug and had no toxicity data collected. Therefore, the adverse event data are based on the 42 patients, who had favorable bio-distribution on imaging dose and received the study treatment.
Arm/Group | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/6 | 15/48
Serious Adverse Events (participants affected / at risk) | 5/5 | 20/37
Other Adverse Events (participants affected / at risk) | 5/5 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg (N=5) | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg (N=37)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Failure to engraft (Investigations) | 0 (0) | 2 (2)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow cellularity (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 2 (3)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 4 (8)
Edema (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 1 (1)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Endocrine - Other (Specify, __) (Endocrine disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 2 (2)
Herpes Zoster (COH) (Infections and infestations) | 1 (1) | 0 (0)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 (0) | 2 (2) — Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 1 (1)
Infection, Fungal (COH) (Infections and infestations) | 0 (0) | 1 (1)
Infection, Viral (COH) (Infections and infestations) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neurology - Other (Specify, __) (Nervous system disorders) | 0 (0) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Investigations) | 2 (2) | 8 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin 1000 cGy + VP-16 40 mg/kg + Cytoxan 100 mg/kg (N=5) | Zevalin 1000 cGy + VP-16 60 mg/kg + Cytoxan 100 mg/kg (N=37)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 4 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 7 (7)
Allergy/Immunology - Other (Specify, __) (Immune system disorders) | 0 (0) | 1 (1)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Failure to engraft (Investigations) | 0 (0) | 2 (2)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (1) | 14 (15)
Bone marrow cellularity (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) | 37 (40)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3) | 6 (6)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 5 (5) | 36 (37)
Lymphopenia (Blood and lymphatic system disorders) | 5 (10) | 37 (46)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3) | 13 (14)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 5 (5) | 35 (35)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 5 (5) | 37 (37)
Transfusion: Platelets (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 5 (5) | 32 (32)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 4 (4) | 30 (30)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 16 (20)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 2 (4)
Hypertension (Cardiac disorders) | 2 (3) | 5 (10)
Hypotension (Cardiac disorders) | 3 (3) | 22 (22)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 5 (9)
Edema (Cardiac disorders) | 3 (3) | 10 (10)
Prothrombin Time (Vascular disorders) | 1 (1) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Vascular disorders) | 2 (2) | 6 (6)
PTT (Partial Thromboplastin Time) (Vascular disorders) | 2 (2) | 4 (4)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 0 (0) | 4 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (6) | 35 (37)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 11 (12)
Insomnia (General disorders) | 4 (4) | 26 (28)
Rigors/chills (General disorders) | 3 (3) | 21 (21)
Sweating (diaphoresis) (General disorders) | 1 (1) | 6 (6)
Weight gain (General disorders) | 0 (0) | 6 (6)
Weight loss (General disorders) | 2 (3) | 12 (12)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (12)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 15 (15)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 16 (17)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 0 (0) | 16 (16)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Rash/desquamation associated with graft versus host disease (GVHD) (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (9) — Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol.
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Endocrine - Other (Specify, __) (Endocrine disorders) | 0 (0) | 2 (2)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (3) | 26 (26)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 10 (10)
Dehydration (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 30 (32)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 11 (11)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 19 (19)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 0 (0) | 5 (5)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 23 (23)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 36 (38)
Salivary gland changes/saliva (Gastrointestinal disorders) | 0 (0) | 7 (7)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 3 (3) | 37 (37)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 13 (13)
Ulcer, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 36 (37)
Hematemesis (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 12 (12)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Melena/GI bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rectal bleeding/hematochezia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hemorrhage, GU (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 0 (0) | 10 (10)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2) | 8 (8)
Hepatic enlargement (Hepatobiliary disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 2 (2) | 30 (30) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1) | 2 (2)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 11 (14)
Herpes Zoster (COH) (Infections and infestations) | 2 (2) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 9 (9) — Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 2 (2)
Infection without neutropenia (Infections and infestations) | 3 (6) | 10 (11)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 2 (2)
Infection, Fungal (COH) (Infections and infestations) | 0 (0) | 1 (1)
Infection, Viral (COH) (Infections and infestations) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (5) | 27 (28)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (5) | 24 (25)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (5) | 37 (37)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Amylase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1) | 26 (26)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (5) | 36 (36)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 4 (4) | 24 (24)
Creatinine (Metabolism and nutrition disorders) | 3 (4) | 10 (10)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (6) | 25 (25)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2) | 9 (9)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (4) | 22 (22)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (5) | 28 (29)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4) | 33 (35)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (4) | 29 (29)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 6 (7)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 0 (0) | 15 (15)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 4 (4)
Hallucinations (Nervous system disorders) | 1 (2) | 4 (5)
Mood alteration (Nervous system disorders) | 4 (5) | 21 (33)
Neurology - Other (Specify, __) (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 12 (13)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 5 (5)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Ocular surface disease (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 0 (0) | 2 (2)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (15) | 32 (88)
Pain - Other (Specify, __) (General disorders) | 2 (3) | 23 (55)
Pneumonia, Other (COH) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 21 (21)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 10 (10)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (14)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (9)
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (12)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine color change (Renal and urinary disorders) | 0 (0) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Investigations) | 2 (2) | 9 (13)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Libido (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Syndromes - Other (Specify, __) (General disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT00562978/Prot_SAP_000.pdf